CLINICAL TRIAL: NCT01500928
Title: Performance Study of the SOLO 2.0 Insulin Pump
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medingo Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTR-135; VTR-075
Record Dates: First submitted 2011-12-11; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Pump; Glycemic Control; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SOLO insulin pump — Use of the SOLO insulin pump for treatment of type 1 diabetes.

SUMMARY:
The Purpose of the study is to to evaluate the performance of the SOLO (version 2.0) micropump insulin delivery system, in Type 1 diabetic patients who use insulin pumps for their treatment.

DETAILED DESCRIPTION:
This is a multi center, one arm, open label and prospective study to assess the safety and quality of the SOLO 2.0 MicroPump Insulin Delivery System, following changes that were done to the SOLO previous version which was validated in 54 subjects.

SOLO 2.0 has the same intended use and core technology as previous SOLO with addition of safety measures, GUI changes and design changes for manufacturability.

The study will include a 30 days treatment period with the Solo MicroPump with no special care required for maintaining glycemic control and with an optional extension period of up to three month in Israel and up to six month in Austria.

The study includes 3 scheduled treatment and one follow up phone call one week after termination of the study. In case of participating the extension period, additional visits will consist once a month.

The study includes 3 scheduled treatment visits and one scheduled telephone call

Visit 1 includes eligibility, baseline evaluation and training in handling of the SOLO System. If no additional practice is required patients will be enrolled. Visit 2 will commence and Solo pump will be filled with insulin. If additional practice is required subject will be sent home for an additional training period of a few days practice using saline and then return for visit 2.

Treatment visits will take place at 3, 10 and 30 days after the enrolment. Additional visits will take place at 60, 90, 120 and 150 days depending on the extension period.

Medical assessment includes DTSQ information, Subject Diary, urine & blood sampling, physical examination, the SOLO Performance Questionnaire, R&D Questionnaire and Complaint Report Forms.Subjects will be asked to record blood glucose measurements, daily activities and carbohydrate consumptions between visits.

Seven days after termination of study treatment a telephone contact with the study subject will take place for the purpose of adverse event reporting and the completion of DTSQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age range:
* 16 to 65 years (Graz)
* 18 to 65 years (Israel)
* Diabetic insulin pump user with diagnosis duration of more than 6 months.
* Subjects who are using Humalog®, NovoRapid®/NovoLog or Apidra® 100U/ml in- - Measures glucose at least four times per day.
* No more than one severe hypoglycemic or ketoacidosis episode within one year
* Willing to sign an informed consent.
* Cooperative, willing to attend all study visits

Exclusion Criteria:

* A1c >= 10.0%
* Two or more documented events of severe hypoglycemia within the previous 12 months
* Diabetes related hospitalization over the past 12 months
* Current significant diabetes-related complications
* Pregnant, lactating or planning to become pregnant during the course of the study
* Substance or alcohol abuse
* Uncontrolled hypertension
* Known dermal hypersensitivity to medical adhesive
* Recurrent episodes of skin infections or dermatological allergies
* Serious or unstable medical or psychological conditions
* Current participation in other clinical studies.
* Working for a competitor company

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Device related safety issues | with in the first month of use
  Subject complaints documented in the R&D questionnaire and Complaint Report Forms which were assessed and found to be device related safety issues.
SOLO use errors | within the first month of use
  Use errors or potential use errors reported in Subject Diary which may be related to SOLO safety.
Device-related adverse outcome | within the first month of use
  Device-related adverse outcome, such as significant skin irritation or infection at the attachment site

SECONDARY OUTCOMES:
Diabetes-related adverse outcome | with in first month of use
  Diabetes-related adverse outcome. i.e. hypoglycemia, hyperglycemia and diabetic ketoacidosis (DKA) events.
Satisfaction iwth SOLO | within the first month of use
  Subject satisfaction with SOLO as reported in:
  1. SOLO performance questionnaire
  2. DTSQ analysis
Product quality (MTBF) | within the first month of use
  Product quality will be assessed by Mean Time Between Failures (MTBF) calculation that include three types of failure modes:
  Type 1: Non-functional device Type 2: Dysfunction that can be recovered by the subject Type 3: Minor issues reported by the user

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, MD, Principal Investigator — Medical University of Graz
Locations (2):
- Israel (2):
  - Schneider Medical Center, Petah Tikva
  - Sourasky Medical Center,, Tel Aviv